CLINICAL TRIAL: NCT00383474
Title: A Phase I Dose-Escalation Study of R115777 (Tipifarnib) Plus PS-341 (Bortezomib) in Relapsed or Refractory Acute Leukemias
Brief Title: Tipifarnib and Bortezomib in Treating Patients With Acute Leukemia or Chronic Myelogenous Leukemia in Blast Phase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00147; NCI-2009-00147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000502258; MCC-14796 (Other: Moffitt Cancer Center); 7306 (Other: CTEP); N01CM62208 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Blastic Phase; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Disease; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Bortezomib; tipifarnib

ARMS (1):
- Arm I (Experimental): Patients will receive an infusion of bortezomib twice a week for 2 weeks. They will also receive tipifarnib by mouth twice a day for 2 weeks.
  Interventions: Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Drug: Tipifarnib

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tipifarnib — Given orally
  Other Names: R115777; Zarnestra

SUMMARY:
This phase I trial is studying the side effects and best dose of tipifarnib and bortezomib in treating patients with acute leukemia or chronic myelogenous leukemia in blast phase. Tipifarnib and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving tipifarnib together with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the dose-limiting toxicity and maximum tolerated dose of tipifarnib and bortezomib in patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, or chronic myeloid leukemia in blast phase.

SECONDARY OBJECTIVES:

I. Determine the effect of this regimen on farnesyltransferase and proteasome inhibition in peripheral blood mononuclear cells in these patients.

II. Determine the clinical efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and oral tipifarnib twice daily on days 1-14. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may continue therapy beyond 6 courses at the discretion of the investigator.

Cohorts of 3-6 patients receive escalating doses of bortezomib and tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood is collected periodically for protein expression studies. Bone marrow aspirates obtained at baseline are examined by immunohistochemistry for Ki-67 activity.

ELIGIBILITY:
Inclusion Criteria:

* Meets 1 of the following disease-specific criteria:

  * Relapsed disease after =< 2 prior chemotherapy regimens (consolidation therapy excluded)
  * Primary-induction failure
  * Previously untreated and deemed unfit for or refusing cytotoxic chemotherapy
* No hyperleukocytosis (leukemic blasts >= 30,000/mm^3)
* No acute promyelocytic leukemia (M3)
* No active CNS leukemia
* SGOT and SGPT =< 2 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine =< 1.5 times ULN
* No uncontrolled hypertension, congestive heart failure, angina pectoris, or ventricular dysrhythmias
* Not pregnant or nursing
* Negative pregnancy test
* No uncontrolled disseminated intravascular coagulation
* Fertile patients must use effective contraception

  * Hormonal contraception must have been initiated ≥ 1 month prior to study entry
* No active graft-vs-host disease
* No active uncontrolled infection
* No intrinsic impaired organ function
* No known allergy to imidazole drugs
* No neuropathy >= grade 1
* No known hypersensitivity to bortezomib, tipifarnib, boron, or mannitol
* No physical or psychiatric conditions that would preclude study participation, including poorly controlled psychosis
* At least 48 hours since prior hydroxyurea
* No prior tipifarnib, bortezomib, or investigational proteasomal inhibitors
* No concurrent radiotherapy, chemotherapy, or immunotherapy
* No concurrent enzyme-inducing antiepileptic medications (e.g., phenytoin, phenobarbital, or carbamazepine)
* ECOG performance status 0-2
* LVEF >= 40%
* Pathologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Chronic myelogenous leukemia in blast phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose of tipifarnib and bortezomib | 21 days

SECONDARY OUTCOMES:
Changes in apoptotic protein expression (Bim, Bax, AKT) | Baseline and day 8
Clinical efficacy (response rate) evaluated using the revised International Working Group Criteria (IWG) for AML | Up to 3 years
Farnesytransferase and proteasome inhibition in peripheral blood mononuclear cells | Day 8
Farnesytransferase and proteasome inhibition in peripheral blood mononuclear cells | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States